CLINICAL TRIAL: NCT04338399
Title: The BURAN Study of Buparlisib (AN2025) In Combination With Paclitaxel Compared to Paclitaxel Alone, in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: The BURAN Study of Buparlisib in Patients With Recurrent or Metastatic HNSCC
Acronym: BURAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Adlai Nortye Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AN2025H0301
Record Dates: First submitted 2020-03-18; First posted 2020-04-08 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Cancer
Keywords: Buparlisib; PD1; PDL1
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — NVP-BKM120; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Buparlisib & Weekly Paclitaxel (Experimental): Drug: Patients will receive 100 mg (2 x 50 mg) buparlisib hard gel capsule administered orally, once daily starting on Day 1 of Treatment Cycle 1, Drug: Paclitaxel (80 mg/m2) administered intravenously (IV) on Days 1, 8, and 15 of a 21-day treatment cycle.
  Treatment will continue until disease progression, unacceptable toxicity, death or discontinuation for any other reason.
- Weekly Paclitaxel (Active Comparator): Patients will receive weekly paclitaxel (80 mg/m2) administered intravenously (IV) on Days 1, 8, and 15 of a 21-day treatment cycle. Treatment will continue until disease progression, unacceptable toxicity, death or discontinuation for any other reason.
  Interventions: Drug: Buparlisib & Paclitaxel

INTERVENTIONS:
Drug: Buparlisib & Paclitaxel — Investigation drug plus paclitaxel
  Other Names: AN2025
  Arms: Weekly Paclitaxel

SUMMARY:
The BURAN study is a randomized, open-label phase III study to assess the treatment effect of once-daily buparlisib in combination with weekly paclitaxel compared to weekly paclitaxel alone in patients with refractory, recurrent, or metastatic head and neck squamous cell carcinoma (HNSCC) that have progressed after prior anti PD 1/anti PD L1 monotherapy; prior anti PD 1/anti PD L1 therapy in combination with platinum-based therapy; or after sequential treatment of anti PD 1/anti PD L1 therapy, either prior to or post, platinum-based therapy.

DETAILED DESCRIPTION:
This study is to assess the impact on overall survival of the combination of Buparlisib and paclitaxel compared to paclitaxel alone in patients with prior anti PD 1/anti PD L1 monotherapy; prior anti PD 1/anti PD L1 therapy in combination with platinum-based therapy; or after sequential treatment of anti PD 1/anti PD L1 therapy, either prior to or post, platinum-based therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years old.
2. Able to provide informed consent obtained before any trial related activities and according to local guidelines.
3. Patient has histologically and/or cytologically-confirmed HNSCC.
4. Patient has archival or new tumor tissue for the analysis of biomarkers and confirmation of HPV status (if unknown). One tumor block (preferred) or a recommended minimum of 5 unstained slides for patients with known HPV status (for tumor DNA characterization) or a recommended minimum of 10 slides for patients whose HPV status is unknown (5 slides for HPV testing plus 5 slides needed for biomarker testing). Enrollment in the study is contingent on confirmation of the availability of an adequate amount of tumor tissue, except in rare special circumstances, which must be reviewed and approved by the sponsor.
5. Patient has either progressive or recurrent disease after treatment with PDL1/PD1 based therapy for recurrent or metastatic disease:

   1. PDLl/PD1 therapy alone for metastatic (monotherapy) disease
   2. PDL1/PD1 in combination with chemotherapy for metastatic and recurrent disease
   3. PDL1/PD1 used for metastatic disease, after or prior to receiving a platinum agent for locally advanced or metastatic disease.
6. 6. Patient has received no more than two prior lines of systemic treatment for HNSCC (single agent chemotherapy used as a radiosensitizer is not counted as a prior line of therapy).
7. Patient has measurable disease as determined per RECIST version 1.1. If the only site of measurable disease is a previously irradiated lesion, documented progression of disease and a four-week period since radiotherapy completion is required.
8. Patient has adequate bone marrow function and organ function as shown by the following:

   1. Absolute neutrophil count (ANC) ≥1.5 x 109/L.
   2. Hemoglobin ≥9 g/dL (which may be reached by transfusion).
   3. Platelets ≥100 x 109/L (which may be reached by transfusion).
   4. International normalized ratio (INR) ≤1.5.
   5. Calcium (corrected for serum albumin) within normal limits (WNL) or ≤ grade 1 severity according to NCI-CTCAE version 5.0 if judged clinically not significant by the Investigator.

      Patients concomitantly taking bisphosphonates or denosumab for calcium correction are eligible.
   6. Normal potassium and magnesium levels.
   7. Alanine aminotransferase (AST) and aspartate aminotransferase (ALT) ≤ 1.5 x upper limit of normal (ULN) or < 3.0 x ULN if liver metastases are present.
   8. Total serum bilirubin ≤ ULN or ≤ 1.5 x ULN if liver metastases are present; or total bilirubin ≤ 3.0 x ULN with direct bilirubin below or within normal range in patients with well documented Gilbert's Syndrome. Gilbert's syndrome is defined as presence of episodes of unconjugated hyperbilirubinemia with normal results from cells blood count (including normal reticulocyte count and blood smear), normal liver function test results, and absence of other contributing disease processes at the time of diagnosis.
   9. Serum creatinine ≤ 1.5 x ULN or calculated and directly measured creatinine clearance (CrCL) > 30 mL/min.
   10. Haemoglobin A1c (glycosylated hemoglobin; HbA1c) ≤8%.
9. Patient has Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
10. Patient is able to swallow and retain oral medication. Patients able to swallow oral medication but mostly self-nourished through gastric or jejunal feeding tube are eligible.
11. Patients must apply highly effective contraception during and throughout the study, as well after the final dose of study treatment

Exclusion Criteria:

Patients meeting any of the following criteria will not be eligible for participation in the study:

1. Patient has received previous treatment with any protein kinase B (PKB/AKT), mammalian target of rapamycin (mTOR) inhibitors, or phosphatidylinositol 3 kinase (PI3K) pathway inhibitors.
2. Patient received treatment with a taxane as part of prior treatment for metastatic disease.
3. Patient has symptomatic central nervous system (CNS) metastases. Patients with asymptomatic CNS metastases may participate in this study. Patient must have completed any prior local treatment for CNS metastases ≥ 28 days prior to the start of study treatment (including radiotherapy) and must be on a stable low dose of corticosteroid therapy. Radiosurgery must have been completed at least 14 days prior to start of study treatment.
4. Patient has received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study treatment or who have adverse events which have not recovered to grade 1 or better from previous chemotherapy treatment (except alopecia, autoimmune endocrine events must be stable and controlled).
5. Patient has grade ≥ 2 neuropathy, colitis, pneumonitis, , and uncontrolled endocrinopathies (e.g., hypothyroidism, diabetes with hemoglobin A1c > 8%) from previous treatment
6. Patient has had major surgery within 14 days prior to starting study treatment or has not recovered from major side effects.
7. Patient is currently receiving increasing or chronic treatment (>5 days) with corticosteroids or another immunosuppressive agent. The following uses of corticosteroids are permitted: single doses; standard premedication for paclitaxel, topical applications (e.g., rash), inhaled sprays (e.g., obstructive airways diseases), eye drops, or local injections (e.g., intra-articular), or < 10 mg prednisolone or equivalent.
8. Patient is being treated at start of study treatment with any of the following drugs:

   1. Drugs known to be strong or moderate inhibitors or inducers of isoenzyme cytochrome P450 3A4 (CYP3A4) including herbal medications (see Table 16).
   2. Drugs with a known risk of inducing Torsades de Pointes. Note: The patient must have discontinued strong inducers for at least one week and must have discontinued strong inhibitors before the treatment is initiated. Switching to a different medication prior to starting study treatment is allowed.
9. Patient is currently receiving warfarin or other coumarin-derived anti-coagulant, for treatment, prophylaxis, or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), fondaparinux or new oral anticoagulants (NOACs) is allowed.
10. Patient has a known hypersensitivity and/or contraindication to paclitaxel, standard premedication for paclitaxel, or other products containing Cremophor®.
11. Patient has other concurrent severe and/or uncontrolled medical conditions that would, in the Investigator's judgment, contraindicate patient participation in the clinical study (e.g., active or uncontrolled severe infection, chronic active hepatitis, immunocompromised, acute or chronic pancreatitis, uncontrolled high blood pressure, interstitial lung disease, etc).
12. Patient has a known history of human immunodeficiency virus (HIV) infection (testing not mandatory).
13. Patient has any of the following cardiac abnormalities:

    1. Symptomatic congestive heart failure within 12 months of the screening period.
    2. History of documented congestive heart failure (New York Heart Association functional classification III-IV) or documented cardiomyopathy and left ventricular ejection fraction (LVEF) <50% as determined by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO).
    3. Myocardial infarction ≤six months prior to enrollment.
    4. Unstable angina pectoris.
    5. Serious uncontrolled cardiac arrhythmia.
    6. Symptomatic pericarditis.
    7. QT interval corrected according to the formula of Fridericia (QTcF) > 450 msec for males and > 470 msec for females, on the screening electrocardiogram (ECG).
    8. Currently receiving treatment with medication that has a known risk to prolong the QT interval or inducing Torsades de Pointes, and the treatment cannot be discontinued or switched to a different medication prior to starting study treatment.
14. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study treatment (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
15. Patient has a medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (e.g., risk of doing harm to self or others), or active severe personality disorders (defined according to the Diagnostic and Statistical Manual of Mental Disorders Fifth Edition [DSM-V]) are not eligible. Note: For patients with psychotropic treatments ongoing at baseline, the dose and the schedule should not be modified within the previous six weeks prior to start of study treatment.
16. Patient has other prior or concurrent malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, or other adequately treated in situ cancer, early gastric or GI cancer resected completely by endoscopy procedures or any other cancer from which the patient has been disease free for ≥ 3years.
17. Patient has a history of non-compliance to any medical regimen or inability to grant consent.
18. Patient is concurrently using or has used another approved or investigational cancer agent within 4 weeks of randomization.
19. Patient is pregnant or nursing (lactating). Patients with elevated human chorionic gonadotrophin (hCG) at baseline that is judged to be related to the tumor are eligible if hCG levels do not show the expected doubling when repeated five to seven days later, or pregnancy has been ruled out by vaginal ultrasound.
20. Patient has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (eg, Flu-Mist®) are live attenuated vaccines, and are not allowed. Non-live COVID vaccinations or boosters should not occur within 30 days of study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 487 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2025-11-02 (Actual); Study Completion 2025-11-02 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Overall survival will be measured from time of randomization until death from any cause. The analysis will occur when all patients have been randomized and followed for 12 months.
  To assess the OS of buparlisib in combination with paclitaxel compared to paclitaxel alone in patients with recurrent or metastatic HNSCC

SECONDARY OUTCOMES:
Progression free survival | PFS will be assessed up to 24 months after all patients are randomized
  Defined as the time from randomization date until tumor progression or death from any cause.
Overall Response Rate | ORR will be assessed for all patients 6 months after randomization is complete.
  Defined at the proportion of patients with a complete or partial response
Health Related Quality of Life (QoL): Time to Definitive deterioration of Quality of Life as assessed by EORTC C30 questionnaire | Assessments will be made from randomization until treatment discontinuation
  A summary of EORTC-QLQ-C30 scores by time window. Time to deterioration is the number of days between the date of randomization and the date of the assessment when definitive deterioration is seen. Definitive deterioration is defined as a decrease in the sub scale score by at least 10% compared with baseline.
Safety and Tolerability of Buparlisib in combination with Paclitaxel compared with Paclitaxel alone as Measured by Number of Participants Experiencing Adverse Events (AEs). | From screening until 4 weeks following treatment discontinuation
  Treatment Emergent Adverse Events AEs will be assessed according to the NCI-CTCAE version 5.0 for severity and will be recorded and classified on the basis of MedDRA terminology.
  Anxiety score change from baseline taken at time of screening (General Anxiety Disorder 7 item scale) until end of treatment.
  Depression score change from baseline taken at time of screening (Patient Health Questionnaire 9) until end of treatment.
Pharmacokinetics of Buparlisib: plasma concentration-time profile of Buparlisib during 15 days of treatment | Day 0 to Day 15 sparse sampling
  For Sparse PK sampling, blood samples will be collected on Treatment Cycle 1, Days 1, 8, and 15 at pre-dose, 1 (± 0.25), 2 ± (0.25) and 6 ± (0.5) hours post-dose. PK sampling will be collected only for those patients randomized to the buparlisib in combination with paclitaxel arm and pharmacokinetic profile of Buparlisib combined with paclitaxel in the study population will be compared with a simulated population PK model.

CONTACTS AND LOCATIONS:
Overall Officials: Senior Director, Global Operations, Study Director — Adlai Nortye USA Inc.
Locations (162):
- United States (21):
  - City of Hope, Duarte, California
  - Yale University, Yale Cancer Center, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Langone, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Cancer Center, Cincinnati, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Hollings Cancer Center, Charleston, South Carolina
  - West Cancer Center, Germantown, Tennessee
  - Hope Cancer Center, UT Health East Texas, Tyler, Texas
- Argentina (6):
  - Fundacion Cenit para la Investigacion en Neurociencias, Buenos Aires
  - Centro de Investigacion Pergamino SA - Clinica Pergamino S.A., Buenos Aires
  - Instituto de Investigaciones Metabólicas (IDIM) // Instituto de Investigaciones Metabólicas S.A., Ciudad Autonoma de Buenos Aire
  - IONC SRL- Instituto Oncológico de Córdoba, Córdoba
  - Fundacion CORI para la Investigacion y Prevencion del Cáncer, La Rioja
  - Centro para la Atencion Integral del Paciente Oncologico - CAIPO, San Miguel de Tucumán
- Princess Alexandra Hospital, Brisbane, Australia
- Belgium (4):
  - Universitair Ziekenhuis Gent UZ Gent, Ghent
  - Universitair Ziekenhuis Brussel, Jette
  - Clinique CHC MontLégia, Liège
  - Clinique Saint-Pierre dOttignies CSPO, Ottignies
- Canada (2):
  - CHUM, Montreal
  - CancerCare Manitoba, Winnipeg
- China (18):
  - Beijing Tongren Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Hunan Cancer Hospital, Changsha
  - Xiangya Hospital Central South University, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - Affiliated Cancer Hospital of Chongqing University, Chongqing
  - The First Affiliated Hospital of CQMU, Chongqing
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Affiliated Cancer Hospital of Guangzhou Medical University, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Anhui Provincial Cancer Hospital, Hefei
  - Shandong Provincial Tumor Hospital, Jinan
  - Yunnan Cancer Hospital, Kunming
  - Cancer Hospital affiliated to Guangxi Medical University, Naning
  - Shanghai Dongfang Hospital, Shanghai
  - Tianjin Cancer Hospital, Tianjin
  - Henan Cancer Hospital, Zhengzhou
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai
- France (12):
  - Centre hospitalier Universitaire de Bordeaux, Bordeaux
  - Centre Franois Baclesse, Caen
  - Centre Leon Berard, Lyon
  - Hopital de la Timone, Marseille
  - Institut regional du Cancer de Montpellier, Montpellier
  - LHopital prive du Confluent Nantes, Nantes
  - Clinique Hartmann, Neuilly-sur-Seine
  - Hôpital St-Louis, Paris
  - Hopital La Pitie Salpetriere, Paris
  - Hopital Tenon, Paris
  - CHP Saint-Grégoire, Saint-Grégoire
  - Institut de cancerologie de Lorraine, Vandœuvre-lès-Nancy
- Germany (11):
  - Uniklinik RWTH Aachen, Aachen
  - Universitaetsklinikum Bonn, Bonn
  - University Hospital Essen, Essen
  - Franziskus Hospital, Georgsmarienhütte
  - HNO-Klinik des Universitats-Klinikums Giessen, Giessen
  - Universitatsmedizin Greifswald - KoR, Greifswald
  - Universitatsklinikum Hamburg Eppendorf, Hamburg
  - Marienkrankenhaus Hamburg, Hamburg
  - Hannover Medical School, Hanover
  - Universitatsklinikum Leipzig, Leipzig
  - UNIVERSITÄTSMEDIZIN Mainz III. Klinik/Poliklinik, Mainz
- Queen Mary Hospital, Hong Kong, Hong Kong
- Hungary (3):
  - Orszagos Onkologiai Intezet, Budapest
  - University of Pecs Department of Oncotherapy, Pécs
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
- Italy (20):
  - Azienda Ospedaliera Universitaria S.Orsola-Malpighi, Bologna
  - ASST Spedali Civili Brescia, Brescia
  - Istituto di Candiolo IRCCS, Candiolo
  - IRCCS - Istituto Scientifico Romagnolo per la Cura e lo Studio dei Tumori, Cesena
  - A.O. S. Croce e Carle, Cuneo
  - Azienda Ospedaliero Universitaria Careggi - Firenze, Florence
  - Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliera San Paolo Polo Universitario, Milan
  - INT IRCCS Fondazione G.Pascale, Napoli
  - A.O.U. "Maggiore della Carita"- S.C.D.U Oncologiac, Novara
  - Azienda Ospedaliero Universitaria Policlinico "Paolo Giaccone" U.O.C. Oncologia Medica, Palermo
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - IRCCS Maugeri Pavia, Pavia
  - IRCCS Istituto Clinico Humanitas, Rozzano
  - AOU San Giovanni di Dio e Ruggi D'Aragona, Università degli Studi di Salerno, Salerno
  - Azienda Ospedaliera Universitaria Senese Policlinico Le Scotte, Siena
  - ASST Valtellina e Alto Lario - UOC Oncologia Medica Ospedale di Sondrio, Sondrio
  - AO Card. G. Panico, Tricase
  - Azienda Sanitaria Universitaria Integrata di Udine, Udine
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Japan (14):
  - Hyogo Cancer Center, Akashi-shi
  - National Cancer Center Hospital, Chūōku
  - Kyushu University Hospital, Fukuoka
  - Saitama Medical University International Medical Center, Hidaka
  - Kagawa University Hospital, Kita-gun
  - Kobe University Hospital, Kobe
  - The Cancer Institute Hospital of JFCR, Kōtoku
  - National Hospital Organization Shikoku Cancer Center, Matsuyama
  - Aichi Cancer Center, Nagoya
  - Kindai University Hospital, Osaka Sayama-shi
  - Hokkaido University Hospital, Sapporo
  - National University Corporation Tohoku University, Tohoku University Hospital, Sendai
  - Showa University Hospital, Shinagawa-Ku
  - Shizuoka Cancer Center, Shizuoka
- Poland (2):
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie, Gliwice
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie, Warsaw
- South Korea (8):
  - Kosin University Gospel Hospital, Busan
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea Seoul ST. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ajou University Hospital, Suwon
- Spain (27):
  - Fundacion Oncologico de Galicia Jos Antonio Quiroga y Pieyro, A Coruña
  - Institut Catala d Oncologia Badalona, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Vall dHebron Institute of Oncology (VHIO), Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Reina Sofia, Córdoba
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital Duran i Reynals - Institut Catala dOncologia ICO, L'Hospitalet de Llobregat
  - Hospital Universitario Severo Ochoa, Leganés
  - Hospital Universitario Lucus Augusti, Lugo
  - Clinica Universidad de Navarra, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca, Madrid
  - Hospital General Universitario Gregorio Maran, Madrid
  - Hospital Puerta de Hierro- Majadahonda, Majadahonda
  - Hospital Regional de Malaga, Málaga
  - Hospital de Navarra, Pamplona
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Santiago de Compostela, Santiago de Compostela
  - Valme Hospital Medical Oncology Department, Seville
  - Instituto Valenciano de Oncologia, Valencia
  - Hospital Clinico Universitario Valencia - INCLIVA, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (7):
  - Changhua Christian Hospital, Changhua
  - Chang Gung Memorial Hospital-KaohSiung, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center Liouying, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital-LinKou, Taoyuan District
- United Kingdom (5):
  - Edinburgh Cancer Center, Edinburgh
  - Beatson Oncology Centre, Glasgow
  - University College London Hospitals, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust - Sutton, Sutton

IPD SHARING:
Plan to Share IPD: No